CLINICAL TRIAL: NCT05337839
Title: Effects of Supervised Versus Unsupervised Home Exercises on Fall-related Variables for Community-dwelling Older Adults
Brief Title: Home Exercises for Fall-related Variables in Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Taciser Kaya, Professor, MD, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21102021TK
Record Dates: First submitted 2022-04-01; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Community-dwelling Older Adults

STUDY DESIGN:
Intervention Model Description: Seventy-five person all of whom eligible and willing were allocated to "supervised home exercise" group (group 1) or "home exercise" group (group 2) using blocked randomisation method. Subjects who have not agreed to join the supervised home exercise group were not invited to join the home exercise group or vice versa.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were informed that they will be requested to do stretching, balance and strengthening exercises. None of the participants did know about the presence of another supervised/unsupervised group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-dwelling older adults receiving supervision (Experimental): Group I; supervised home exercise group
  Interventions: Procedure: home exercises
- Community-dwelling older adults not supervised (Active Comparator): Group II; unsupervised home exercise group
  Interventions: Procedure: home exercises

INTERVENTIONS:
Procedure: home exercises — stretching, balance and strengthening exercises

SUMMARY:
The aim was to measure and compare the effects of supervised and unsupervised home exercises on the fall related variables.

DETAILED DESCRIPTION:
There are several studies investigating the beneficial effects of exercise on physical function among elderly. However the trials that reporting beneficial effects of an exercise programme on psychosocial functions such as depression and falls efficacy are scarcend. And also these trials are designed to compare fully supervised experimental group with a control group receiving usual care. In only one, out of these studies, supervision was minimal and delivered via home visit. However no psychosocial function related outcome measure was evaluated. In the present study the investigators have intended to assess the effects of minimally supervised home exercise programme on physical and psychosocial fall related variables by comparing with unsupervised home exercise programme in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform timed up and go (TUG) test
* not having regular exercise habit
* a score above 20 on the Mini Mental State Examination (MMSE)

Exclusion Criteria:

* medical conditions impeding to perform exercises such as severe musculoskeletal and neurological disease, severe visual impairment, cardiovascular, pulmonary or malignant disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-02-20 (Actual); Primary Completion 2013-07-20 (Actual); Study Completion 2013-10-20 (Actual)

PRIMARY OUTCOMES:
Falls efficacy | baseline, eighth week, sixth month
  It was assessed using the Falls Efficacy Scale International (FES-I). FES-I is a self-rating questionnaire designed for measuring concerns about the possibility of falling during several activities of daily living. In total, sixteen practices and activities, which are carried out at home such as cooking, dressing, taking a bath; and out of home such as visiting someone, walking on an uneven surface or shopping are scored between 1 and 4 (1 = not at all concerned, 4 = very concerned). The range of total score varies between 16 to 64 and the higher the score the lower the falls efficacy. The investigators have aimed to measure the change in falls efficacy between three time points (baseline, eighth week, sixth month)in order to explore whether there is an improvement in this outcome measure. The change in falls efficacy was calculated by using suitable nonparametric statistical analysis methods.

SECONDARY OUTCOMES:
Fear of Falling (FOF) | baseline, eighth week, sixth month
  Visual Analog Scale (VAS) was used for measuring FOF subjectively. Participants were asked to indicate the degree of falling fear by making a mark on a 100 milimeter line (zero; not at all, 100; maximum fear). A new paper sheet was used at each visit so that the participants couldn't see the previous response that they have given. This was done with the purpose of prevent them from getting biased.
Functional Mobility | baseline, eighth week, sixth month
  To assess functional mobility Timed up and go (TUG) test was used. Participants were requested to walk at their ordinary walking speed during TUG test. They were seated at the beginning of the test and asked for rising from chair after the command "ready-set-go", walking 3 meters, turning around, going back to chair and sitting down again. Duration between rising from chair and sitting down was recorded with a stopwatch. Before testing, participants were instructed about testing procedure and one test trial was performed for this purpose.
Balance Performance | baseline, eighth week, sixth month
  With the aim of rating balance performance, Balance Performance Oriented Mobility Assessment (BPOMA) of Tinetti was used. In this test, eight different tasks are scored between 0-2. Maximum possible score is 16 and higher score is related to the better balance performance. For detailed information; this test evaluates sitting and standing balance, turning 360°, the ability of arising from chair and sitting down.
Fall risk | baseline, eighth week, sixth month
  Elderly Falls Screening Test (EFST) was used to assess risk of fall. It is composed of two parts, one of which queries fall number in the last year, history of injurious fall and near fall; the second evaluates walking speed and style. The first part is self-report and covers three items; the second part is scored by assessor and covers two items. Maximum possible score is five. A score between 0-1 indicates low, 2-3 moderate and 4-5 high fall risk.
Geriatric Depression Scale Short Form (GDS-SF) | baseline, eighth week, sixth month
  This scale is used for defining the depressive symptoms. It covers fifteen dichotomous questions that ask participants to answer in a yes or no fashion. Of the 15 questions, 10 indicate the presence of depression when answered as yes while remaining five indicate the presence of depression when answered as no. An answer in the direction of depression is assumed as one point. To get a final score, all points are summed. Thus, total score is between 0-15. A score between 0-5 is normal, a score above 5 suggests depression.

CONTACTS AND LOCATIONS:
Overall Officials: Taciser Kaya, Prof., MD, Principal Investigator — Izmir Bozyaka Training and Reseach Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjerk M, Brovold T, Skelton DA, Bergland A. A falls prevention programme to improve quality of life, physical function and falls efficacy in older people receiving home help services: study protocol for a randomised controlled trial. BMC Health Serv Res. 2017 Aug 14;17(1):559. doi: 10.1186/s12913-017-2516-5. PMID 28806904
- [Background] Lacroix A, Kressig RW, Muehlbauer T, Gschwind YJ, Pfenninger B, Bruegger O, Granacher U. Effects of a Supervised versus an Unsupervised Combined Balance and Strength Training Program on Balance and Muscle Power in Healthy Older Adults: A Randomized Controlled Trial. Gerontology. 2016;62(3):275-88. doi: 10.1159/000442087. Epub 2015 Dec 9. PMID 26645282
- [Background] Youssef EF, Shanb AA. Supervised Versus Home Exercise Training Programs on Functional Balance in Older Subjects. Malays J Med Sci. 2016 Nov;23(6):83-93. doi: 10.21315/mjms2016.23.6.9. Epub 2016 Dec 7. PMID 28090182
- [Background] Rapp K, Freiberger E, Todd C, Klenk J, Becker C, Denkinger M, Scheidt-Nave C, Fuchs J. Fall incidence in Germany: results of two population-based studies, and comparison of retrospective and prospective falls data collection methods. BMC Geriatr. 2014 Sep 20;14:105. doi: 10.1186/1471-2318-14-105. PMID 25241278
- [Derived] Avci Trakyali A, Kaya T, Ince B. Effects of an exercise program combining unsupervised home exercises and supervised group-based exercises on fall-related variables in older adults: a randomized controlled trial. Eur Geriatr Med. 2023 Feb;14(1):59-67. doi: 10.1007/s41999-022-00724-3. Epub 2022 Dec 14. PMID 36515868